CLINICAL TRIAL: NCT01003873
Title: Effect of Weight Loss Induced Either by Gastric Bypass or Lifestyle Intervention on the Peripheral Activity of the Endocannabinoid System
Brief Title: Gastric Bypass and Peripheral Activity of the Endocannabinoid System
Acronym: CCENDO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2008/19
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Obesity
Keywords: morbid obesity; bariatric surgery; lifestyle intervention; endocannabinoids system
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy of visceral and peripheral adipose tissue will be done during surgery and peripheral adipose tissue will be done 6 months after surgery
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bypass gastric: First arm is represented by obese patients that will be studied before and after a gastric bypass. They will be studied before surgery as well as 1 month and 6 months after surgery.
  Interventions: Biological: Evaluation of the endocannabinoid system; Procedure: Biopsy of visceral and peripheral adipose tissue; Biological: Evaluation of metabolic parameters; Behavioral: Evolution of behavioral parameters; Behavioral: Dietician consultation; Behavioral: Psychologist consultation
- Lifestyle intervention: The second group is represented by obese patients that will be studied before lifestyle intervention, 6 months after the beginning of the intervention and after a time that will allow patients to lose the same amount of weight that patients that had been through surgery had lost one month after surgery.
  Interventions: Biological: Evaluation of the endocannabinoid system; Biological: Evaluation of metabolic parameters; Behavioral: Evolution of behavioral parameters; Behavioral: Dietician consultation; Behavioral: Psychologist consultation
- Control subjects: The third group is a control group of normal weight people that will be studied at one time and after 6 months with stable weight.
  Interventions: Biological: Evaluation of the endocannabinoid system; Biological: Evaluation of metabolic parameters; Behavioral: Evolution of behavioral parameters

INTERVENTIONS:
Biological: Evaluation of the endocannabinoid system — The evaluation of the endocannabinoid system consist in the determination of plasma concentration of the 2 main endocannabinoids (2AG and AEA) before (5 blood samples) and after (5 blood samples) after consumption of a calibrated food. As a comparator, ghrelin will be measured at the same time.
Procedure: Biopsy of visceral and peripheral adipose tissue — The endocannabinoids will be also determined in adipose tissue. Biopsy of visceral and peripheral adipose tissue will be done during surgery and peripheral adipose tissue will be done 6 months after surgery.
  Groups: Bypass gastric
Biological: Evaluation of metabolic parameters — The evaluation of the metabolic status consist in evaluation of body composition (DEXA), determination of visceral adiposity (CT scan) and measurement of plasma lipids, glucose, insulin, leptin, adiponectin.
Behavioral: Evolution of behavioral parameters — The behavioral evaluation will de done with different questionnaires: ORWELL 97, HAD scale, Three Factor Eating Questionnaire, Beck Depression inventory, Questionnaire of personality TCI.
Behavioral: Dietician consultation — The evaluation of the metabolic status will also be seen by a dietician.
  Groups: Bypass gastric; Lifestyle intervention
Behavioral: Psychologist consultation — The behavioural evaluation will de done with a psychologist consultation
  Groups: Bypass gastric; Lifestyle intervention

SUMMARY:
The aim of the study is to precise the effect of a large amount of weight loss induced by gastric bypass on the endocannabinoid system (plasma and adipose tissue) of morbidly obese patients and to determine the influence of a gastric bypass surgery compared to a lifestyle intervention with equivalent weight loss on the endocannabinoid system

DETAILED DESCRIPTION:
Dysregulation of the endocannabinoid system has been associated with the development of obesity, metabolic and cardiovascular disorders in both animals and humans.

Obese patients, especially those with abdominal obesity, have significantly higher levels of endocannabinoids. No influence of moderate (5%) body weight loss (induced either by diet intervention or sibutramine) on the peripheral activity of the endocannabinoid system gastric bypass (GB) surgery is the most efficient treatment of obesity Hormonal pathways may participate to the weight reducing effect of the procedure.The endocannabinoid system is present in the gastrointestinal tract.

In animals, sustained weight loss after GB is characterized by reduction of endocannabinoids levels.

The endocannabinoid levels will be studied (baseline and after stimulation) in:

* Normal-weight subjects
* Obese subjects before and after gastric bypass surgery
* Obese subjects before and after a lifestyle intervention

ELIGIBILITY:
Inclusion Criteria:

* Arms 1 and 2:
* Age between 18 and 60
* BMI > 40kg/m² or at least 30kg/m² with complication
* Medical follow up before surgery
* Patients that engaged themselves to a long medical follow up
* Efficient contraception
* Written, informed consent of each subject before the beginning of the study
* Arm 3:
* Age between 18 and 60
* BMI between 18 and 25 kg/m²
* Stable weight over the 3 past months
* Restrain score <4 disinhibition <6and hunger > 4 at the TFEQ
* No job in the endocrinology department
* Written, informed consent of each subject before the beginning of the study

Exclusion Criteria:

* Arms 1,2 and 3
* No care of obesity before inclusion
* Incapacity of the patient to follow a medical follow up
* Drug or alcohol abuse
* Urine test result positive for THC
* Threaten life diseases
* Pregnancy, breast feeding
* Smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 2 groups : from primary care clinic
  * obese patients with gastric bypass
  * obese patients with lifestyle intervention 1 group : volunteer
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2009-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Plasmatic endocannabinoïd concentration variation | Inclusion and 6 month-follow up

SECONDARY OUTCOMES:
Plasma concentration of the endocannabinoids during food exposure | At each visit
Post prandial pic of the plasma concentration of the endocannabinoids | At each visit
Adipose tissue concentration of the endocannabinoids | Inclusion and 6 month-follow up
Plasma concentration of adipokines | At each visit
Body mass index | At each visit
Body composition | At each visit
Insulin sensitivity | At each visit
Area under the curve of plasma concentration of 2AG | Inclusion and 6 month follow-up
Questionaries scores | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Blandine GATTA-CHERIFI, MD, Principal Investigator — University Hospital, Bordeaux, France; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux, France
Locations (1):
- Haut Lévêque Hospital, Endocrine department, Pessac, France

REFERENCES:
- [Background] Di Marzo V, Matias I. Endocannabinoid control of food intake and energy balance. Nat Neurosci. 2005 May;8(5):585-9. doi: 10.1038/nn1457. PMID 15856067
- [Background] Cota D. CB1 receptors: emerging evidence for central and peripheral mechanisms that regulate energy balance, metabolism, and cardiovascular health. Diabetes Metab Res Rev. 2007 Oct;23(7):507-17. doi: 10.1002/dmrr.764. PMID 17683024
- [Background] Engeli S, Bohnke J, Feldpausch M, Gorzelniak K, Janke J, Batkai S, Pacher P, Harvey-White J, Luft FC, Sharma AM, Jordan J. Activation of the peripheral endocannabinoid system in human obesity. Diabetes. 2005 Oct;54(10):2838-43. doi: 10.2337/diabetes.54.10.2838. PMID 16186383
- [Background] Bluher M, Engeli S, Kloting N, Berndt J, Fasshauer M, Batkai S, Pacher P, Schon MR, Jordan J, Stumvoll M. Dysregulation of the peripheral and adipose tissue endocannabinoid system in human abdominal obesity. Diabetes. 2006 Nov;55(11):3053-60. doi: 10.2337/db06-0812. PMID 17065342
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408